CLINICAL TRIAL: NCT05681507
Title: Efficacy of Transversus Thoracic Muscle Plane Block in Adult Cardiac Surgery: A Randomized Controlled Trial
Brief Title: Efficacy of TTMPB in Adult Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eric Albrecht (Other)
Responsible Party: Sponsor-Investigator, Eric Albrecht, Professor of Clinical Anesthesia, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TTMPB-Heart Trial (2022-01126)
Record Dates: First submitted 2022-12-13; First posted 2023-01-12 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Acute Post Operative Pain
Keywords: Transversus Thoracic Muscle Plane Block; Adult Cardiac Surgery; Sternotomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Patients will benefit of our institutional intensive-care unit analgesia protocol
  Interventions: Procedure: Standard postoperative analgesia
- Intervention group (Experimental): Patients will benefit of a transversus thoracic muscle plane block and our institutional intensive-care unit analgesia protocol
  Interventions: Drug: Transversus thoracic muscle plane block

INTERVENTIONS:
Drug: Transversus thoracic muscle plane block — Ultrasound guided bilateral parasternal injection of bupivacain 0.375%, 20ml, at 4th thoracic vertebral level.
  Other Names: TTMPB
  Arms: Intervention group
Procedure: Standard postoperative analgesia — Standard of postoperative ICU analgesic care, per institutional protocol
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to compare the efficacy of Transversus Thoracic Muscle Plane Block (TTMPB) integrated in a modern multimodal analgesia protocol, following the ERAS® recommendations, in adult patients undergoing planned open heart surgery.

The main study question is:

Does the addition of TTMPB to a standard analgesic protocol significantly improve analgesia following elective open heart surgery?

The investigators will primarily compare postoperative opioid consumption and pain scores in patients who will be randomly allocated to one of two groups:

The control group will receive standard analgesia per institutional Intensive Care Unit protocol.

The intervention group will receive the same standard of care plus a TTMP block (40ml of bupivacaine 0.375%, total dose of 150 mg).

The investigators will also study the impact of group allocation on secondary outcomes, such as the rate of early mobilization.

ELIGIBILITY:
Inclusion Criteria:

* Direct informed consent as documented by signature
* Major adult (≥ 18 years old) with body weight ≥ 50 kg. For the record, fifty kilograms is the minimal weight to ensure that participants remain safely away from maximal doses of LA (3 mg/kg)
* Planned and primary cardiac surgery via a sternotomy approach
* Planned for ultra-fast-track procedure (i.e. postoperative extubation time of maximum two hours)

Exclusion Criteria:

* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Refusal and/or inability to understand or sign the informed consent
* Emergent cardiac surgery
* Previous cardiac surgery
* Known hypersensitivity or true allergy to bupivacaine and other amide-class LA
* Chronic pain history
* Substance abuse history
* Inability to follow the procedures of the study (e.g. due to language problems, psychological / psychiatric disorders, dementia)
* Clinically significant concomitant diseases: severe cardiac dysfunction (i.e. LVEF ≤ 35%); severe chronic obstructive pulmonary disease (i.e. FEV < 50%); severe hepatic disease.
* Severe obesity (BMI > 35kg/m2)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Total amount (in mg) of opioid consumption within the first 24 hours | 24 hours
  Total opioid consumption

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Rancati, Attending physician, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- CHUVaudois, Lausanne, Canton of Vaud, Switzerland